CLINICAL TRIAL: NCT02891174
Title: A Randomized-controlled Trial to Assess the Effect of Ibuprofen on Post-partum Blood Pressure in Women With Hypertensive Disorders of Pregnancy
Brief Title: The Effect of Ibuprofen on Post-partum Blood Pressure in Women With Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elizabeth Langen, Assistant Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00117154
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Hypertension, Pregnancy-Induced; Pre-eclampsia
Keywords: ibuprofen; acetaminophen; blood pressure; post-partum; pain control; pre-eclampsia; gestational hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Agnosia | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen followed by acetaminophen (Active Comparator): Ibuprofen administered immediately post-partum, 600 mg (3 x 200 mg tablets) every 6 hours for 24 hours followed by acetaminophen, 650 mg (2 x 325 mg tablets) every 6 hours for 24 hours.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen
- Acetaminophen followed by ibuprofen (Active Comparator): Acetaminophen administered immediately post-partum, 650 mg (2 x 325 mg tablets) every 6 hours for 24 hours followed by ibuprofen, 600 mg (3 x 200 mg tablets) every 6 hours for 24 hours.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — At the time of delivery, eligibility will be reviewed. If the participant remains eligible, she will be randomized by the study pharmacy to begin post-partum analgesic therapy with ibuprofen followed by acetaminophen.
  Other Names: Advil; Motrin
Drug: Acetaminophen — At the time of delivery, eligibility will be reviewed. If the participant remains eligible, she will be randomized by the study pharmacy to begin post-partum analgesic therapy with acetaminophen followed by ibuprofen.
  Other Names: Tylenol

SUMMARY:
To assess the effect of routine doses of ibuprofen on post-partum blood pressure control in women with gestational hypertension (gHTN) or preeclampsia without severe features (preE).

DETAILED DESCRIPTION:
Non-steroidal anti-inflammatory drugs (NSAIDs) are frequently prescribed for post-partum analgesia. This use is supported by limited data on post-partum pain specifically; however, ibuprofen and other NSAIDs are superior to acetaminophen in ameliorating uterine pain and cramping in dysmenorrhea. The effect of NSAIDs on blood pressure (BP) in women post-partum is less well-known. In non-pregnant hypertensive patients NSAIDs are associated with increased BP over short courses of days to months, though effects of various NSAIDs differ. Pooled analyses suggest changes in mean BP of up to 3-6 mm Hg depending on the measurement method.There are case reports of hypertensive crises after NSAID administration post-partum in both normotensive and hypertensive women. A larger, recent retrospective cohort study found no difference in mean arterial pressure (MAP) or need for antihypertensive therapy in women with severe hypertensive disorders of pregnancy who were exposed to NSAIDs post-partum.

In light of the potential for worsening blood pressure in women with hypertensive disorders of pregnancy, the Task Force on Hypertension in Pregnancy of American College of Obstetricians and Gynecologists stated that "providers should be reminded of the contribution of nonsteroidal anti-inflammatory agents to increased BP." Additionally the task force recommends that NSAIDS "be replaced by other analgesics in women with hypertension that persists for more than 1 day postpartum". However, provider practices since the publication of these guidelines have varied.

Hypothesis: When compared to acetaminophen, ibuprofen does not increase post-partum systolic blood pressure (SBP) above baseline to a clinically relevant degree (≥10 mmHg) in women with gHTN and preE.

Aim 1: To assess the mean difference in SBP during 24 hours of exposure to ibuprofen and acetaminophen.

Aim 2: To assess whether ibuprofen results in higher satisfaction with pain control in the immediate post-partum period (48 hours) compared to acetaminophen.

Aim 3: To prospectively assess the need for post-partum anti-hypertensive therapy and readmission for blood pressure control in women with gHTN and preE. The post-partum period is defined as delivery through 6 weeks after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Antepartum women
* Diagnosis of Gestational Hypertension or Pre-eclampsia by blood pressure ≥140 systolic or ≥90 diastolic, on at least 2 measurements ≥ 4 hours apart; with or without proteinuria (urine protein-creatinine ratio ≥0.3 or 24 hour-urine protein ≥300 mg).
* Taking one or fewer oral medications for blood pressure control.
* Singleton gestation.
* English-speaking

Exclusion Criteria:

* Allergy to nonsteroidal anti-inflammatory drugs, aspirin, or acetaminophen
* More than 1 severe range blood pressure (≥160 systolic or ≥110 diastolic) prior to enrollment.
* Neurologic symptoms attributed to hypertension (headache, visual changes) prior to enrollment.
* Pulmonary edema.
* Elevated AST (>60 international units/L) or ALT (>70 international units/L) prior to enrollment.
* Low platelet count (<100,000/microliter) prior to enrollment.
* Renal insufficiency (creatinine > 1.1 or double the baseline creatinine if known) prior to enrollment.
* Chronic hypertension defined as hypertension pre-existing pregnancy or diagnosed prior to 20-weeks' gestation.
* Moderate- or severe-persistent asthma.
* Therapeutic anticoagulation.
* Chronic opiate use during the pregnancy (opiate therapy given daily for > 2 weeks).
* Lactose intolerance or allergy due to placebo containing lactose.
* Cesarean delivery.
* Additional anesthesia at time of delivery (spinal anesthesia, sedation) that would change routine pain management.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jourdan Triebwasser, MD, Principal Investigator — University of Michigan; Elizabeth Langen, MD, Principal Investigator — University of Michigan; Alexander Tsodikov, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 women were consented prior to delivery.
  Women were subsequently excluded due to cesarean delivery (n=20), severe features of preeclampsia (n=7), additional anesthesia (n=2), and delivery physician preference (n=2).
  43 women were randomized. Six women declined study medication and were not included in intention-to-treat analysis.
Groups:
- Ibuprofen Followed by Acetaminophen: Period 1: Ibuprofen 600 mg every 6 hours for 24 hours Period 2: Acetaminophen 650 mg every 6 hours for 24 hours. No washout
- Acetaminophen Followed by Ibuprofen: Period 1: Acetaminophen 650 mg every 6 hours for 24 hours Period 2: Ibuprofen 600 mg every 6 hours for 24 hours. No washout
Period: First Intervention (24 Hours)
Arm/Group | Ibuprofen Followed by Acetaminophen | Acetaminophen Followed by Ibuprofen
Started | 20 | 23
Received First Intervention | 19 | 18
Completed | 17 | 10
Not Completed | 3 | 13
Not completed — Declined any study medication | 1 | 5
Not completed — Discharged prior to cross-over | 0 | 2
Not completed — Withdrew after receiving study drug | 2 | 6
Period: Second Intervention (24 Hours)
Arm/Group | Ibuprofen Followed by Acetaminophen | Acetaminophen Followed by Ibuprofen
Started | 17 | 10
Completed | 11 | 3
Not Completed | 6 | 7
Not completed — No blood pressure after cross-over | 1 | 0
Not completed — Discharged during second intervention | 3 | 5
Not completed — Withdrew after receiving study drug | 2 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were measured after the first milestone, after 6 total participants who were initially randomized declined the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen Followed by Acetaminophen | Acetaminophen Followed by Ibuprofen | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (6.9) | 31.1 (6.3) | 31.0 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 17 | 17 | 34
  Race/Ethnicity: Black | 1 | 0 | 1
  Race/Ethnicity: Hispanic | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 33.5 [30 to 41] | 31.7 [28 to 36] | 32.3 [29.2 to 36.9]
Marital Status [Count of Participants; unit: Participants]
  Single | 4 | 5 | 9
  Lives with partner | 1 | 1 | 2
  Married | 14 | 11 | 25
  Not reported | 0 | 1 | 1
Insurance [Count of Participants; unit: Participants]
  Commercial | 17 | 14 | 31
  Public/Medicaid | 2 | 4 | 6
Nulliparous [Count of Participants; unit: Participants] | 10 | 11 | 21
Gestational Age [Mean (Standard Deviation); unit: weeks] | 39.4 (1.5) | 38.6 (1.5) | 38.9 (1.5)
Gestational Hypertension [Count of Participants; unit: Participants] | 15 | 17 | 32
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 132.5 (5.3) | 131.2 (7.3) | 131.6 (10.9)
Maximum Systolic Blood Pressure Prior to Delivery [Mean (Standard Deviation); unit: mmHg] — The maximum systolic blood pressure between admission and delivery for each participant was recorded. The mean of the maximum systolic blood pressures was calculated for each group.
  mmHg | 153.2 (8.8) | 149.8 (8.6) | 151.5 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Systolic Blood Pressure (SBP)
Description: The adjusted mean difference in systolic blood pressure after 24 hours of exposure each to ibuprofen and acetaminophen.
Time Frame: 24 hours following intervention
Population: 37 women who received >=1 dose of study drug were included in intention-to-treat analyses. 35 women had blood pressure recorded in the intended ibuprofen period; 2 excluded due to discharge prior to cross-over. 36 women had blood pressure recorded in the intended acetaminophen period; 1 excluded with no blood pressure measured after cross-over.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Ibuprofen: Intention to treat population: received at least 1 dose of study medication in the first intervention period (either ibuprofen or acetaminophen), and had a blood pressure measured during the intended ibuprofen period.
- Acetaminophen: Intention to treat population: received at least 1 dose of study medication in the first intervention period (either ibuprofen or acetaminophen), and had a blood pressure measured during the intended acetaminophen period.
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 35 | 36
mmHg
  Baseline systolic blood pressure | 131.8 (6.3) | 132.0 (6.4)
  Systolic blood pressure after exposure | 129.1 (8.3) | 129.1 (8.5)
  Observed Difference in systolic blood pressure | -2.7 (8.1) | -2.9 (8.6)
Statistical Analysis 1: Comparison: Ibuprofen vs Acetaminophen; Test type: Equivalence — margin=10 mmHg; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-3.7 to 5.7] — The adjusted mean difference between ibuprofen and acetaminophen is presented here. The adjusted mean difference was calculated using a linear mixed model adjusting for time period by intention-to-treat principles

2. Secondary Outcome: Change in Self-reported Pain Score 2 Hours After First Intervention
Description: Prior to the first dose of pain medication, participants will take a brief, self-administered survey to assess abdominal and overall pain using a 0-10 scale. Two hours after the first dose of study drug, participants will repeat the self-administered survey to assess abdominal, perineal, and overall pain using a 0-10 scale. Clinical Pain Scale: 0=no pain to 10=worst pain.
Time Frame: At the time of first dose of study drug and 2 hours after
Population: 14 women in the ibuprofen first group and 8 women in the the acetaminophen first group completed pain surveys before and 2 hours after 1st dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ibuprofen: Ibuprofen was the first intervention and pain scales were administered only during this first period.
- Acetaminophen: Acetaminophen was the first intervention and pain scales were administered only during this first period.
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 14 | 8
score on a scale
  Abdominal pain | -0.6 (1.6) | -0.3 (1.2)
  Perineal pain | -1.1 (1.6) | 1.0 (0.6)
  Overall pain | -0.7 (1.8) | -0.6 (0.9)
Statistical Analysis 1: Comparison: Ibuprofen vs Acetaminophen; Change in abdominal pain; Test type: Superiority; p = 0.59, t-test, 2 sided — Abdominal pain
Statistical Analysis 2: Comparison: Ibuprofen vs Acetaminophen; Change in perineal pain; Test type: Superiority; p = 0.91, t-test, 2 sided — Perineal pain
Statistical Analysis 3: Comparison: Ibuprofen vs Acetaminophen; Change in overall pain; Test type: Superiority; p = 0.88, t-test, 2 sided — Overall pain

3. Secondary Outcome: Mean Pain Score by Nursing Assessment
Description: Pain scores using a 0-10 scale as assessed by nursing during the 48 hours from initial study medication administration will be abstracted from the participant's medical record. Clinical Pain Scale: 0=no pain to 10=worst pain. All pain scores during the first intervention (0-24 hours) and second intervention (24-48) are included according to intention-to-treat principles.
Time Frame: 0-24 hours and 24-48 hours after initial study medication administration
Population: Of 37 women in intention-to-treat analyses, 35 were analyzed in ibuprofen treatment; 2 of those women had no recorded nursing pain score in ibuprofen period (n=33). 36 women were analyzed in acetaminophen treatment, but 1 of those women had no recorded nursing pain score in acetaminophen period (n=35).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen | Acetaminophen
Number analyzed (Participants) | 33 | 35
score on a scale | 2.2 (1.1) | 2.3 (1.3)
Statistical Analysis 1: Comparison: Ibuprofen vs Acetaminophen; Test type: Other; p = 0.76, t-test, 2 sided

4. Secondary Outcome: Satisfaction With Pain Control During 24 Hours of Exposure Each to Ibuprofen and Acetaminophen
Description: A brief survey on satisfaction with pain control during the first 24 hours post-partum and the second 24 hours post-partum, as well as overall during post-partum stay will be administered prior to discharge using a 1-5 Likert scale: 1=not satisfied to 5=extremely satisfied.
Time Frame: 24 hours and 48 hours after initial study medication administration
Population: 11 women in the ibuprofen first group and 6 women in the the acetaminophen first group completed the satisfaction survey prior to discharge.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Ibuprofen Followed by Acetaminophen: Period 1: Ibuprofen 600 mg every 6 hours for 24 hours. Period 2: Acetaminophen 650 mg every 6 hours for 24 hours. No washout period.
- Acetaminophen Followed by Ibuprofen: Period 1: Acetaminophen 650 mg every 6 hours for 24 hours. Period 2: Ibuprofen 600 mg every 6 hours for 24 hours. No washout period.
Arm/Group | Ibuprofen Followed by Acetaminophen | Acetaminophen Followed by Ibuprofen
Number analyzed (Participants) | 11 | 6
units on a scale
  Period 1 | 3 [2 to 4] | 4 [4 to 5]
  Period 2 | 3 [2 to 4] | 4.5 [4 to 5]
  Overall | 3 [2 to 4] | 4.5 [4 to 5]
Statistical Analysis 1: Comparison: Ibuprofen Followed by Acetaminophen vs Acetaminophen Followed by Ibuprofen; First intervention (24 hours); Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Ibuprofen Followed by Acetaminophen vs Acetaminophen Followed by Ibuprofen; Second intervention (24 hours); Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ibuprofen Followed by Acetaminophen; Overall satisfaction with pain control during study period; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 48 hours
Groups:
- Ibuprofen: Women who received ibuprofen intervention
- Acetaminophen: Women who received acetaminophen intervention
Arm/Group | Ibuprofen | Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/34
Other Adverse Events (participants affected / at risk) | 0/29 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02891174/Prot_SAP_000.pdf